CLINICAL TRIAL: NCT05154357
Title: The Effect Of Elastic Sac On Physıological Characteristic And Feeding Performance In Preterm Infants
Brief Title: The Effect of Elastic Sac on Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Canan Uzun, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: E-74555795-050.01.04-88001
Record Dates: First submitted 2021-11-05; First posted 2021-12-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Oxygen Saturation; Heart Rate; Nutritional Status
Keywords: Heart rate; Oxygen Saturation; Preterm Infants; Safe Swaddling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Half an hour before the first feeding hour, the infant's heart rate and oxygen saturation will be recorded. Then, he/she will be placed in the elastic sac, positioned and will be allowed to take a rest until the feeding hour for 30 minutes. His/her physiological parameters will be recorded ten minutes before the feeding time, during feeding and ten minutes after feeding. When the feeding time begins, the chronometer will be started and it will be stopped when feeding is completed. At the second feeding time, the infant's heart rate and oxygen saturation will be recorded half an hour before the feeding hour. Then, he/she will be positioned without performing any different application and will be allowed to take a rest until the feeding time. His/her physiological parameters will be recorded ten minutes before the feeding time, during feeding and ten minutes after feeding. When feeding begins, the chronometer will be started and when it is over, the chronometer will be stopped.
  Interventions: Other: Elastic Sac; Other: Control
- Group 2 (Experimental): Half an hour before the first feeding time of the infant, his/her heart rate and oxygen saturation will be recorded. Then, he/she will be positioned without performing any different application and will be allowed to take a rest until the feeding time. His/her physiological parameters will be recorded ten minutes before the feeding hour, during feeding and ten minutes after feeding. When feeding begins, the chronometer will be started and when it is over, the chronometer will be stopped. At the second feeding hour, the infant's heart rate and oxygen saturation will be recorded half an hour before the feeding hour. Then, he/she will be placed in the elastic sac, positioned, and allowed to take a rest until the feeding hour. His/her physiological parameters will be recorded ten minutes before the feeding hour, during feeding and ten minutes after feeding. When feeding begins, the chronometer will be started and when it is over, the chronometer will be stopped.
  Interventions: Other: Elastic Sac; Other: Control

INTERVENTIONS:
Other: Elastic Sac — Half an hour before the feeding time, the infant will be placed in the elastic sac, be laid in the right lateral position within the nest with an angle of 45 degrees and will be allowed to take a rest within the elastic sac for half an hour. At the feeding time, he/she will be fed by the researcher with a bottle in the right lateral position within the elastic sac with an angle of 45 degrees without making any change in his/her position.
Other: Control — Half an hour before the feeding time, the infant will be laid in the right lateral position within the nest with an angle of 45 degrees without performing any different application and will be allowed to take a rest. At the feeding time, he/she will be fed by the researcher with a bottle in the right lateral position within the elastic sac with an angle of 45 degrees without making any change in his/her position.

SUMMARY:
The study will be conducted using the crossover randomized controlled method. Preterm infants who began oral feeding from the neonatal intensive care unit will be divided into two groups through randomization in the computer environment. Following the randomization, infants in Group 1 will be fed by applying ''elastic sac'' at the first feeding hour after they are included in the study and in the next feeding they will be fed without performing any application. Infants in Group 2 will be fed without performing any application at the first feeding hour after they are included in the study and they will be fed at the second feeding hour by applying ''elastic sac''. Infants in both groups will be fed by the researcher with a bottle in a semi-fowler right lateral position during feeding hours. During feeding, the effect of the elastic sac on the infant's feeding status and physiological parameters will be evaluated.

DETAILED DESCRIPTION:
Swaddling method is a method which can be used for preserving thermoregulation, decreasing stress and maintaining comfort in term and preterm infants during painful procedures. The effect of the ''elastic sac'' method which is thought to imitate the uterus environment, on physiological parameters and feeding performance of infants during feeding will be evaluated. The ''elastic sac'' method will be applied with 100% cotton and elastic fabric. The single-use elastic and cotton fabric was sewed as a U-shaped sac for each infant included in the study. The infant will be placed in the sac during the feeding hour and will be placed in a position in which he/she can move easily, maintain the flexion posture and feel safe contrary to traditional swaddling. The purpose of the study is to evaluate stress-associated physiological parameters and feeding status during oral feeding in preterm infants starting oral feeding. The study will be conducted using the crossover randomized controlled method. The sample size of the study was determined via the power analysis in accordance with the results obtained from studies conducted via a similar research method. According to the results of the analyses, a total of 26 preterm infants including 13 for each group will be included in the study group. After informing the families of infants meeting the inclusion criteria both in written and oral forms, the study will be conducted with mothers who agree to participate in the study and their infants.

Application Stages GROUP 1

1. Feeding Time Half an hour before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form. The infant will be placed in the ''elastic sac'' and the angle of the incubator bed will be elevated 45 degrees. He/she will be laid in the right lateral position within the nest and will be allowed to take a rest within the ''elastic sac'' until the feeding time (30 minutes). Giving priority to breast milk, formula milk at optimum temperature will be prepared for infants without breast milk. The nutrient amount ordered by the doctor will be put in the bottle. Ten minutes before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form every two minutes. At the feeding time, the bottle will be approached to the infant's mouth for feeding in the semi-fowler right lateral position at 45 degrees without making any change in his/her posture. As soon as the infant begins to suck, the chronometer will be started and the infant's heart rate and oxygen saturation will be recorded by another observer nurse every two minutes throughout feeding. When the infant shows signs of fatigue (Spo2 less than 90, HR higher than 160), the feeding will be discontinued and when the infant's HR fall below 160 and spO2 increases above 90, the feeding will continue. The time of feeding will be limited to a maximum of 30 minutes. When the infant stops feeding, the chronometer will be stopped, the feeding will be terminated and the infant will be allowed to take a rest. His/her heart rate and oxygen saturation will be recorded in the observation form every two minutes for ten minutes. Then, the ''elastic sac'' application will be terminated and an onesie will be put on the infant in line with the care procedures of the clinic and he/she will be allowed to take a rest until the next feeding hour. The amount (cc) of milk the infant receives from the ordered amount of the milk and the amount of nutrient he/she receives in a minute will be calculated and recorded in the observation form.
2. Feeding Time Half an hour before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form. The angle of the incubator bed will be elevated 45 degrees. Only an onesie will be put on the infant in line with the care procedures of the clinic and no other application will be performed. He/she will be laid in the right lateral position within the nest and will be allowed to take a rest until the feeding time. In order to feed him/her the same nutrient at both feeding hours, the same nutrient prepared at the previous feeding hour will be prepared at optimum temperature. The nutrient amount ordered by the doctor will be put in the bottle. Ten minutes before the feeding hour, the infant's heart rate and oxygen saturation will be recorded in the observation form every two minutes. At the feeding hour, the bottle will be approached to the infant's mouth for feeding in the semi-fowler right lateral position at 45 degrees without making any change in his/her position. As soon as the infant begins to suck, the chronometer will be started and the infant's heart rate and oxygen saturation will be recorded by another observer nurse every two minutes throughout feeding. When the infant shows signs of fatigue (Spo2 less than 90, HR higher than 160), the feeding will be discontinued and when the infant's HR falls below 160 and spO2 increases above 90, the feeding will continue. The time of feeding will be limited to a maximum of 30 minutes. When the infant stops feeding, the chronometer will be stopped, the feeding will be terminated and the infant will be allowed to take a rest. His/her heart rate and oxygen saturation will be recorded in the observation form every two minutes for ten minutes. The infant will be allowed to take a rest in line with the care procedures of the clinic. The amount (cc) of milk the infant receives from the ordered amount of the milk and the amount of nutrient he/she receives in a minute will be calculated and recorded in the observation form.

GROUP 2

1. Feeding Time Half an hour before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form. The angle of the incubator bed will be elevated 45 degrees. Only an onesie will be put on the infant in line with the care procedures of the clinic and no other application will be performed. He/she will be laid in the right lateral position within the nest and will be allowed to take a rest until the feeding time (30 minutes). Giving priority to breast milk, formula milk at optimum temperature will be prepared for infants without breast milk. The nutrient amount ordered by the doctor will be put in the bottle. Ten minutes before the feeding hour, the infant's heart rate and oxygen saturation will be recorded in the observation form every two minutes. At the feeding hour, the bottle will be approached to the infant's mouth for feeding in the semi-fowler right lateral position at 45 degrees without making any change in his/her position. As soon as the infant begins to suck, the chronometer will be started and the infant's heart rate and oxygen saturation will be recorded by another observer nurse every two minutes throughout feeding. When the infant shows signs of fatigue (Spo2 less than 90, HR higher than 160), the feeding will be discontinued and when the infant's HR falls below 160 and spO2 increases above 90, the feeding will continue. The time of feeding will be limited to a maximum of 30 minutes. When the infant stops feeding, the chronometer will be stopped, the feeding will be terminated and the infant will be allowed to take a rest. His/her heart rate and oxygen saturation will be recorded in the observation form every two minutes for ten minutes. The infant will be allowed to take a rest until the next feeding hour in line with the care procedures of the clinic. Amount (cc) of milk the infant receives from the ordered amount of the milk and the amount of nutrient he/she receives in a minute will be calculated and recorded in the record form.
2. Feeding Time Half an hour before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form. The infant will be placed in the ''elastic sac'' and the angle of the incubator bed will be elevated 45 degrees. He/she will be laid in the right lateral position within the nest and will be allowed to take a rest within the elastic sac until the feeding time. In order to feed him/her the same nutrient at both feeding hours, the same nutrient prepared during the previous feeding hour will be prepared at optimum temperature. The nutrient amount ordered by the doctor will be put in the bottle. Ten minutes before the feeding time, the infant's heart rate and oxygen saturation will be recorded in the observation form every two minutes. At the feeding time, the bottle will be approached to the infant's mouth for feeding in the semi-fowler right lateral position at 45 degrees without making any change in his/her position. As soon as the infant begins to suck, the chronometer will be started and the infant's heart rate and oxygen saturation will be recorded by another observer nurse every two minutes throughout feeding. When the infant shows signs of fatigue (Spo2 less than 90, HR higher than 160), the feeding will be discontinued and when the infant's HR falls below 160 and spO2 increases above 90, the feeding will continue. The time of feeding will be limited to a maximum of 30 minutes. When the infant stops feeding, the chronometer will be stopped, the feeding will be terminated and the infant will be allowed to take a rest. His/her heart rate and oxygen saturation will be recorded in the observation form every two minutes for ten minutes. Then, the ''elastic sac'' application will be terminated and he/she will be allowed to take a rest in line with the care procedures of the clinic. The amount (cc) of milk the infant receives from the ordered amount of the milk and the amount of nutrient he/she receives in a minute will be calculated and recorded in the observation form.

ELIGIBILITY:
Criteria Inclusion Criteria

* Parent agreeing to take part in the study
* Infant starting oral feeding by the doctor in the neonatal intensive care unit and tolerating it
* Infant born at 26-36+6 gestational week specified according to the last menstruation date of the mother
* Infant being at 32-39+6 postmenstrual week
* Infant having a body weight of 1500 grams and above
* Infant being fed orally once before and tolerating it
* Infant having no health problem except for being a preterm

Exclusion Criteria

* Infant having a gastrointestinal, neurological or genetic illness (such as necrotizing enterocolitis, intracranial bleeding, hydrocephaly, omophalocele, down's syndrome, gastroschisis) and other illnesses
* Infant having no obstacle to oral feeding (such as cleft palate, cleft lip, facial muscle paralysis, craniofacial anomaly)
* Infant being on oxygen support

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Feeding Status | maximum 30 minutes
  In order to assess the feeding status of the infant, his/her time of feeding and the amount of nutrient he/she receives in a minute will be calculated. In order to determine his/her time of feeding, a phone chronometer will be started as soon as he/she begins feeding and it will be stopped when feeding is over. All infants in Group 1 and Group 2 will be fed with a slow-flow bottle branded Avent which is designed for premature infants. It will be calculated how much (cc) of the total amount of nutrient ordered by the doctor the infant receives. The total amount of nutrient received by the infant will be divided into the time of feeding and thus the amount of nutrient received in a minute (cc) will be calculated.

SECONDARY OUTCOMES:
Heart Rate | All babies in Group 1 and Group 2 will be recorded in the registration form by the observing nurse once half an hour before the feeding time, 10 minutes before the feeding time, during the feeding and at 2-minute intervals 10 minutes after the feeding.
  In order to determine the infant's heart rate, a 'Covidien' pulse oximeter will be used. It will be recorded by the observer nurse in the observation form every two minutes once half an hour before the feeding hour of all infants in Group 1 and Group 2, ten minutes before the feeding hour, throughout feeding and ten minutes after feeding.
Oxygen Saturation | All babies in Group 1 and Group 2 will be recorded in the registration form by the observing nurse once half an hour before the feeding time, 10 minutes before the feeding time, during the feeding and at 2 minutes intervals 10 minutes after the feeding.
  In order to determine the infant's oxygen saturation, a 'Covidien' pulse oximeter will be used. It will be recorded by the observer nurse in the observation form every two minutes once half an hour before the feeding time of all infants in Group 1 and Group 2, ten minutes before the feeding hour, throughout feeding and ten minutes after feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu GÖZEN, Prof., Principal Investigator — Istanbul University - Cerrahpasa; Fatma Narter Kaya, Assoc. Prof., Principal Investigator — Istanbul Dr. Lütfi Kırdar Şehir Hastanesi
Locations (1):
- Istanbul University, Cerrahpaşa, Istanbul, Turkey (Türkiye)